CLINICAL TRIAL: NCT03005912
Title: Clinical Single Centre Cohort Study Comparing Telephone vs. Voice Over Internet Protocol (VoIP) Speech Comprehension for Acoustical and Bluetooth Speech Signal Transmission in Hearing Aided Subjects.
Brief Title: Telephone vs. Voice Over IP Speech Comprehension in Hearing Aided Subjects.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cochlear (Industry); Stiftung Besser Hören (Unknown)
Responsible Party: Principal Investigator, Markus Huth, Oberarzt, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Bluetooth-Study; 2016-01935 (Other: Kantonale Ethikkommission Bern)
Record Dates: First submitted 2016-06-26; First posted 2016-12-30 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Hearing-Impairment
Keywords: Speech Comprehension; Telephony; VoIP
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional acoustic telephony (Placebo Comparator): Telephone speech comprehension in hearing aided patients (Cochlear Implant or GN Resound hearing aid) for a conventional mobile phone call with acoustic transmission of the speech signal.
  Interventions: Device: Conventional acoustic telephony
- Conventional bluetooth telephony (Active Comparator): Telephone speech comprehension in hearing aided patients (Cochlear Implant or GN Resound hearing aid) for a conventional mobile phone call with direct bluetooth transmission of the speech signal to the cochlear implant or hearing aid.
  Interventions: Device: Conventional bluetooth telephony
- VoIP acoustic telephony (Active Comparator): Telephone speech comprehension in hearing aided patients (Cochlear Implant or GN Resound hearing aid) for a VoIP mobile phone call with acoustic transmission of the speech signal.
  Interventions: Device: VoIP acoustic telephony
- VoIP bluetooth telephony (Active Comparator): Telephone speech comprehension in hearing aided patients (Cochlear Implant or GN Resound hearing aid) for a VoIP mobile phone call with direct bluetooth transmission of the speech signal to the cochlear implant or hearing aid.
  Interventions: Device: VoIP bluetooth telephony

INTERVENTIONS:
Device: Conventional acoustic telephony — Quantification of speech comprehension by means of the Hochmair-Schulz-Moser sentence test.
  Arms: Conventional acoustic telephony
Device: Conventional bluetooth telephony — Quantification of speech comprehension by means of the Hochmair-Schulz-Moser sentence test.
  Arms: Conventional bluetooth telephony
Device: VoIP acoustic telephony — Quantification of speech comprehension by means of the Hochmair-Schulz-Moser sentence test.
  Arms: VoIP acoustic telephony
Device: VoIP bluetooth telephony — Quantification of speech comprehension by means of the Hochmair-Schulz-Moser sentence test.
  Arms: VoIP bluetooth telephony

SUMMARY:
Despite modern hearing aids such as cochlear implants, speech comprehension during telephone conversation is challenging for hearing-impaired patients. On the one hand, conventional telephones transmit a limited spectrum of the acoustic signal compared to a normal conversation. On the other hand, lip reading during a phone call is generally not possible. As a result, speech comprehension during a telephone conversation is reduced. In previous studies, the authors demonstrated an improved speech comprehension for hearing-impaired patients using voice-over internet protocol (VoIP) telephony (Skype) compared to conventional telephony.

New bluetooth-enabled hearing aids allow for direct transmission of the telephone signal to the hearing device. As the direct transmission is expected to improve signal-to-noise ratio, speech comprehension is tested in patients with bluetooth-enabled hearing aids for 4 different scenarios: 1. conventional telephony without bluetooth device 2. conventional telephony with bluetooth device 3. VoIP telephony without bluetooth device 4. VoIP telephony with bluetooth device

DETAILED DESCRIPTION:
Speech comprehension of hearing impaired individuals is limited in telephone conversations due to the limited acoustic spectrum transmitted by conventional analogue telephones, such as background noise, interferences with the hearing aid and the absent possibility of lip-reading. This can provide an impact on quality of life as better speech comprehension reduces exclusion from social interactions as well as potential professional occupations. Furthermore, in elderly population an impaired hearing function is associated with a higher risk of dementia, mortality rate and dependency in the daily activities.

Mantokoudis et al. recently demonstrated that the larger acoustic spectrum of internet telephony (Voice over Internet Protocol [VoIP]) results in superior speech comprehension of individuals with hearing aids compared to conventional telephones. Low signal quality during internet telephony does not significantly attenuate speech understanding. Another study revealed that internet telephony combined with a webcam further improves speech comprehension as additional lip reading was possible.

New bluetooth audio streaming devices allow for pairing with smart phones or other devices supporting bluetooth technology such as computers for direct routing of the audio signal to the hearing aid. Current state of research shows significant benefits for hearing impaired individuals using this technology for telephone conversations. The speech comprehension and subjective satisfaction can be improved due to a better sound quality and accuracy and less noise interference.

However, speech comprehension of these new bluetooth devices has not been investigated in combination with internet telephony (VoIP) and it remains unclear whether hearing impaired individuals could benefit of this possibility. This study investigates, whether bluetooth audio streaming devices paired to hearing aids/implants combined with internet telephony improves speech comprehension in hearing impaired individuals.

VoIP and conventional telephone speech comprehension will be compared with and without a wireless bluetooth phone clip (Cochlear Wireless Phone Clip, Cochlear Ltd., 1 University Avenue, Macquarie University, New South Wales 2109, Australia). The phone clip is capable to directly connect to other bluetooth-enabled devices and transmits the audio signal directly to the sound processor of the hearing implant. A microphone in the phone clip enables to record and transmit the user's spoken words to the mobile phone therefore a hands-free use is possible.

Bluetooth connection is a well-established wireless technology transmitting at 2.4 gigahertz at distances up to approximately seven meters. The wireless technology is the same for most of bluetooth and Wireless Local Area Network (WLAN) devices. According to the Swiss federal health office the electromagnetic radiation of the bluetooth device as intended to be used in the proposed study fulfils the requirements of the European Committee for Electrotechnical Standardization (CENELEC).

Several previous studies demonstrated a significantly increased conventional telephone speech perception with the Cochlear Wireless Phone Clip than without this device. On the other hand, speech perception in hearing impaired people using internet telephony is improved compared to conventional telephony. However, speech perception using the phone clip in connection to internet telephony has not been studied to this date and remains unknown.

The purpose of the proposed study is to quantify VoIP vs. conventional telephone speech comprehension in individuals with or without application of bluetooth phone clip. Potentially better speech comprehension due to the application of the phone clip could alleviate the handicap of communication in individuals with hearing aids. As a consequence the social life and contacts of the affected individuals such as worsening of mental state and dependency in the everyday life could be ameliorated only by using a simple device.

The goal of this study is to measure speech comprehension of individuals with hearing aids using a bluetooth paired phone clip and VoIP telephony. To quantify a potential benefit of this, speech comprehension has to be tested with and without the phone clip for VoIP and conventional telephony in the same individuals. Speech comprehension will be quantified with a signal/noise ratio of the HSM- sentence test (Hochmair, Schulz, Moser)

Upon agreement to participate, patients are invited to the audiological department at Inselspital in Bern. After remaining questions are clarified, the patient has to sign a written informed consent. The investigation will take approximately two hours and takes place in the sound-proof hearing test chambers of the audiological department.

Four different speech comprehension scenarios are tested:

1. Conventional telephony without bluetooth device
2. Conventional telephony with bluetooth device
3. VoIP telephony without bluetooth device
4. VoIP telephony with bluetooth device

To evaluate speech comprehension, the HSM (Hochmair-Schulz-Moser) sentence test is used. This is a test mainly applied to evaluate the speech comprehension in patients with cochlear implants and consists of 30 lists each including 20 short sentences. After initial presentation of exercise sentences without background noise, additional noise is added while the speech signal is kept at a constant volume level. The percentage of speech comprehension is determined by the quantity of correctly understood sentences at a certain signal-to-noise ratio (S/N Ratio). In this study a S/N Ratio of 10dB, with a signal at 70dB and noise at 60dB, will be analysed.

For representativeness of speech comprehension results, participants will use their hearing aids with their daily use volume settings. The phone clip will be programmed for a 1:1 transmission of the telephone conversation and the ambient noise. At the end, the patient has to evaluate the subjective perception of the speech sound quality by means of the Mean Opinion Score (MOS).

ELIGIBILITY:
Inclusion Criteria:

* Bluetooth enabled hearing aid (Nucleus 6 CI or a GN Resound hearing aid) compatible to the phone clip
* Use of hearing aid for ≥ 3 months.
* Native German speaker

Exclusion Criteria:

* Mentally or physically unfit to participate
* Vulnerable Person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Speech comprehension scores | 2 years
  Speech comprehension scores of the HSM-sentence test for each patient with and without bluetooth connection will be measured and compared in conventional and internet telephony.

SECONDARY OUTCOMES:
Subjective perception of speech sound quality | 2 years
  Subjective perception of speech sound quality by means of the Mean Opinion Score (MOS).

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Mantokoudis, MD, Principal Investigator — Attending physician
Locations (1):
- University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tyler RS, Baker LJ, Armstrong-Bednall G. Difficulties experienced by hearing-aid candidates and hearing-aid users. Br J Audiol. 1983 Aug;17(3):191-201. doi: 10.3109/03005368309107884. PMID 6357328
- [Background] Cray JW, Allen RL, Stuart A, Hudson S, Layman E, Givens GD. An investigation of telephone use among cochlear implant recipients. Am J Audiol. 2004 Dec;13(2):200-12. doi: 10.1044/1059-0889(2004/025). PMID 15903146
- [Background] Ito J, Nakatake M, Fujita S. Hearing ability by telephone of patients with cochlear implants. Otolaryngol Head Neck Surg. 1999 Dec;121(6):802-4. doi: 10.1053/hn.1999.v121.a93864. PMID 10580241
- [Background] Liu C, Fu QJ, Narayanan SS. Effect of bandwidth extension to telephone speech recognition in cochlear implant users. J Acoust Soc Am. 2009 Feb;125(2):EL77-83. doi: 10.1121/1.3062145. PMID 19206836
- [Background] Horng MJ, Chen HC, Hsu CJ, Fu QJ. Telephone speech perception by Mandarin-speaking cochlear implantees. Ear Hear. 2007 Apr;28(2 Suppl):66S-69S. doi: 10.1097/AUD.0b013e31803153bd. PMID 17496651
- [Background] Fu QJ, Galvin JJ 3rd. Recognition of simulated telephone speech by cochlear implant users. Am J Audiol. 2006 Dec;15(2):127-32. doi: 10.1044/1059-0889(2006/016). PMID 17182877
- [Background] Milchard AJ, Cullington HE. An investigation into the effect of limiting the frequency bandwidth of speech on speech recognition in adult cochlear implant users. Int J Audiol. 2004 Jun;43(6):356-62. doi: 10.1080/14992020400050045. PMID 15457818
- [Background] Kepler LJ, Terry M, Sweetman RH. Telephone usage in the hearing-impaired population. Ear Hear. 1992 Oct;13(5):311-9. doi: 10.1097/00003446-199210000-00009. PMID 1487091
- [Background] Rumeau C, Frere J, Montaut-Verient B, Lion A, Gauchard G, Parietti-Winkler C. Quality of life and audiologic performance through the ability to phone of cochlear implant users. Eur Arch Otorhinolaryngol. 2015 Dec;272(12):3685-92. doi: 10.1007/s00405-014-3448-x. Epub 2014 Dec 20. PMID 25527411
- [Background] Cacciatore F, Napoli C, Abete P, Marciano E, Triassi M, Rengo F. Quality of life determinants and hearing function in an elderly population: Osservatorio Geriatrico Campano Study Group. Gerontology. 1999 Nov-Dec;45(6):323-8. doi: 10.1159/000022113. PMID 10559650
- [Background] Dalton DS, Cruickshanks KJ, Klein BE, Klein R, Wiley TL, Nondahl DM. The impact of hearing loss on quality of life in older adults. Gerontologist. 2003 Oct;43(5):661-8. doi: 10.1093/geront/43.5.661. PMID 14570962
- [Background] Gates GA, Cobb JL, Linn RT, Rees T, Wolf PA, D'Agostino RB. Central auditory dysfunction, cognitive dysfunction, and dementia in older people. Arch Otolaryngol Head Neck Surg. 1996 Feb;122(2):161-7. doi: 10.1001/archotol.1996.01890140047010. PMID 8630210
- [Background] Barnett S, Franks P. Deafness and mortality: analyses of linked data from the National Health Interview Survey and National Death Index. Public Health Rep. 1999 Jul-Aug;114(4):330-6. doi: 10.1093/phr/114.4.330. PMID 10501133
- [Result] Mantokoudis G, Kompis M, Dubach P, Caversaccio M, Senn P. How internet telephony could improve communication for hearing-impaired individuals. Otol Neurotol. 2010 Sep;31(7):1014-21. doi: 10.1097/MAO.0b013e3181ec1d46. PMID 20634771
- [Result] Mantokoudis G, Dubach P, Pfiffner F, Kompis M, Caversaccio M, Senn P. Speech perception benefits of internet versus conventional telephony for hearing-impaired individuals. J Med Internet Res. 2012 Jul 16;14(4):e102. doi: 10.2196/jmir.1818. PMID 22805169
- [Result] Mantokoudis G, Dahler C, Dubach P, Kompis M, Caversaccio MD, Senn P. Internet video telephony allows speech reading by deaf individuals and improves speech perception by cochlear implant users. PLoS One. 2013;8(1):e54770. doi: 10.1371/journal.pone.0054770. Epub 2013 Jan 24. PMID 23359119
- [Result] Wolfe J, Morais M, Schafer E. Improving Hearing Performance in Cochlear Nucleus 6 users with true wireless accessories. Cochlear Limited. 2015 May; D710887 ISS2
- [Result] Robier M, Bakhos D, Pawelczyk T, Lescanne E. Evaluation of benefit provided by the Cochlear Wireless Phone Clip. Cochlear Limited.2015 Dec; D785163 ISS1
- [Result] Martinez Basterra Z, Fernández de Pinedo M, Altuna Mariexcurrena X. Telephone speech recognition improvement in a noisy environment: use of a Bluetooth accessory. Cochlear Limited.2015 Dec; D785163 ISS1
- [Result] Kim MB, Chung WH, Choi J, Hong SH, Cho YS, Park G, Lee S. Effect of a Bluetooth-implemented hearing aid on speech recognition performance: subjective and objective measurement. Ann Otol Rhinol Laryngol. 2014 Jun;123(6):395-401. doi: 10.1177/0003489414526847. PMID 24687593
- [Result] Marcrum SC. Wireless streaming with the Cochlear Wireless Phone Clip improves speech understanding and reduces listening effort during telephone use in noise. Cochlear Limited.2015 Dec; D785163 ISS1
- [Result] Gündüz B, Gökdoğan C, Orçan E, Fikret Çetik M, Tuncer Ü, Özdemiroğlu S. Hearing inventory with the Cochlear Wireless Phone Clip in experienced adult cochlear implant recipients at work and during daily life. Cochlear Limited.2015 Dec; D785163 ISS1
- [Result] Duke M, Wolfe J. Evaluation of speech recognition over the telephone with and without the Cochlear Wireless Phone Clip. Cochlear Limited.2015 Dec; D785163 ISS1
- [Result] Çiprut A, Derinsu U, Cesur S, Çiçek B, Özkan B, Yücel E. Speech intelligibility with the Cochlear Wireless Phone Clip in experienced cochlear implant recipients. Cochlear Limited.2015 Dec; D785163 ISS1
- [Result] Qian H, Loizou PC, Dorman MF. A phone-assistive device based on Bluetooth technology for cochlear implant users. IEEE Trans Neural Syst Rehabil Eng. 2003 Sep;11(3):282-7. doi: 10.1109/TNSRE.2003.816871. PMID 14518792
- [Result] Hochmair-Desoyer I, Schulz E, Moser L, Schmidt M. The HSM sentence test as a tool for evaluating the speech understanding in noise of cochlear implant users. Am J Otol. 1997 Nov;18(6 Suppl):S83. PMID 9391610